CLINICAL TRIAL: NCT06657781
Title: Study and Role of Inflammasome in Platelet Activation During Bacterial And/or Viral Sepsis
Acronym: PLAQSEPSIS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RIPH3_2022/03
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Bacterial Sepsis
Keywords: Sepsis; platelet; NLRP3; BTK; IL-1β
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- leptospirosis: patient suffering from leptospirosis
- bacterial: patient suffering from bacterial infections including in-hospital-acquired-infections
- viral: patient suffering from viral infection except COVID-19
- Control: patients non infected
- viral infection SARS-COv2 +: patient suffering from COVID-19 previously enrolled in PLAQCOVID trial.

SUMMARY:
: Sepsis, now defined as life-threatening organ dysfunction due to a dysregulated host response to infection, is an important global health problem representing about a fifth of all global deaths. It can be associated, in some cases, with multiple organ failure and cytokine storm. The main objective of this study is to estimate and to compare the activation rate of the Nucleotide-binding domain Leucine Rich repeat containing Protein 3 (NLRP3) inflammasome in platelets between five groups of patients suffering from bacterial and/or viral sepsis, with different severity levels according to Sequential Organ Failure Assessment (SOFA) score to precise the platelets' implication in this cytokine storm.

DETAILED DESCRIPTION:
Patients with bacterial or vial sepsis have been shown to exhibit very high levels of pro-inflammatory cytokines (IL1, IL6, IFN, IP10 and MCP1) that may activate the T-helper-1 lymphocytic response (Th1). These cytokines can be produced by several cell types, including blood platelets. IL1 is an important pro-inflammatory cytokine whose expression is increased in various pro-inflammatory contexts, including dengue infection. It induces an increase in endothelial permeability and a pro-thrombotic state, as described in patients infected with COVID-19. It is synthesized as a protein precursor that is cleaved by the NLRP3 (Nucleotide-binding domain Leucine repeat Rich containing Protein 3). Close associations between the deregulation of inflammasome activity and hereditary or acquired diseases suggest an important role of NLRP3 inflammasome in regulating immune responses. The activation of the NLRP3 inflammasome increases caspase 1 activity and induces the production of bioactive IL1 as well as other pro-inflammatory cytokines such as IL18. The major role of NLRP3 platelet inflammasome in the "cytokine storm" has been highlighted in the case of Dengue virus infection. We hypothesize that blood platelets may play an important role in the inflammatory response observed during sepsis through the activation of NLRP3 inflammasome, particularly during its exacerbation.

* Five groups of patients will be constituted: patients with leptospirosis, patients with bacterial infections including in-hospital-acquired-infections, patients with viral infection, patients non infected (control group), patients with viral infection SARS-COv2 +.
* Only one blood collection will be realized

ELIGIBILITY:
Inclusion Criteria:

* For all groups: patients older than 18 years at inclusion and acceptation of participation by the patient, his relative or his legal representative (depending on the situation)
* For groups 1, 2, 3 and 5: Patient with a confirmed sepsis (microbiological confirmation)
* For group 4 : Patient non infected

Exclusion Criteria:

* Refusal of participation by the patient, his relative or his legal representative (depending on the situation)
* Patients subject to a safeguard measure of justice
* Patients younger than 18 years at inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty patients will be included in each group: patients with leptospirosis, patients with bacterial infections including in-hospital-acquired-infections, patients with viral infection, patients non infected (control group).
  Fifty-one patients will be included in group of patients with viral infection SARS-COv2 +.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Nucleotide-binding domain Leucine Rich repeat containing Protein 3 activation | Baseline
  The primary outcome will be the evaluation of platelets' NLRP3 activation in septic patients according to the severity of the disease

SECONDARY OUTCOMES:
Confocal Microscopy | Baseline
  We aim to confirm the colocalization of NRLP3/ASC in inflammasome activation by confocal microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric MARTINO, Doctor, Principal Investigator — chu de pointe à pitre
Locations (1):
- Centre Hospitalier Universitaire de la Guadeloup, Les Abymes, Guadeloupe, Guadeloupe

IPD SHARING:
Plan to Share IPD: No